CLINICAL TRIAL: NCT05048485
Title: Tuberculosis - Learning the Effect of Parasites and Reinforcing Diets (TB-LEOPARD)
Brief Title: Tuberculosis - Learning the Effect of Parasites and Reinforcing Diets
Acronym: TB-LEOPARD
Status: Completed | Type: Observational
Sponsor: Boston Medical Center (Other)
Collaborators: Jawaharlal Institute of Postgraduate Medical Education & Research (Other Government)
Responsible Party: Sponsor
Other Study IDs: H-41912; H-41912 (Other Grant/Funding Number: Burroughs Wellcome)
Record Dates: First submitted 2021-09-09; First posted 2021-09-17 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Tuberculosis, Pulmonary; Helminthiasis; Malnutrition
Keywords: Nutritional supplements; TB LION; India
MeSH Terms: conditions — Tuberculosis, Pulmonary; Helminthiasis; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, sputum and stool samples will be collected and some samples will be retained for future testing. The PaxGene tubes will be collected and stored for future analysis to study RNA sequences for transcriptional differences between persons with TB with and without intestinal infections. Plasma samples and analysis of analytes will be analyzed to investigate further the immunologic mechanisms and to assess how these responses are modulated over time by treatment of parasites and by feeding individuals. Serum samples will be retained for future analysis of micronutrients and assessment of the immune response. Stool samples will be frozen for future microbiome analysis. Sputum samples obtained for the study will be assessed for differentially culturable TB variants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LEOPARD Cohort 1: Control group: The study will enroll 50 newly diagnosed smear-positive (>/=1+ AFB) pulmonary TB patients whose household contacts are enrolled in the TB-LION study and who are not receiving nutritional supplementation.
  TB LION group: The study will enroll 50 newly diagnosed smear-positive (>/=1+ AFB) pulmonary TB patients whose household contacts are enrolled in the TB-LION study and who are receiving nutritional supplementation.
- LEOPARD Cohort 2: The study will enroll 300 newly diagnosed smear-positive (>/=1+ AFB) pulmonary TB patients whose household contacts are not enrolled in the TB-LION study.

SUMMARY:
The objectives of this research are to determine:

* the burden of intestinal parasitic infections among persons living with pulmonary tuberculosis (TB)
* whether intestinal parasitic infections alter TB treatment outcomes, including speed of sputum clearance and treatment outcomes
* the impact of malnutrition on speed of sputum clearance and TB treatment outcomes
* whether nutritional supplementation improves speed of sputum clearance and treatment outcomes

In this study the researchers will investigate how intestinal parasites impact the nutritional status of TB patients before the start of nutritional supplementation and how they alter the trajectory of weight gain in those receiving supplementation by analyzing results from 2 cohorts.

LEOPARD Cohort 1-

* Control-Enroll TB cases, screen for undernutrition, obtain stool for intestinal parasite screening by polymerase chain reaction (PCR), and assess them for treatment outcomes and weight gain
* TB LION (Learning Impact of Nutrition) - Enroll TB cases, provide nutritional supplementation for 6 months (as part of existing TB LION study), screen for undernutrition, obtain stool for intestinal parasite screening by PCR, and assess them for treatment outcomes and weight gain

LEOPARD Cohort 2 -

* Enroll TB cases, screen for undernutrition, obtain stool for internal parasite screening by PCR, and assess them for treatment outcomes and weight gain.

DETAILED DESCRIPTION:
LEOPARD Cohort 1-

Control:

* Pulmonary TB patients who are newly diagnosed smear-positive (>/=1+ Acid-fast bacillus/AFB) and whose household contacts are enrolled in the TB-LION (Learning Impact of Nutrition) study but are not receiving nutritional supplementation
* 50 participants will be enrolled and followed for up to 12 months
* Stool sample will be collected at the week 1 visit (visit 2)
* Blood samples will be collected the screening visit, week 1, month 2, and month 6
* Sputum samples will be collected at the screening visit, week 1, week 2, and month 6

TB LION:

* Pulmonary TB patients who are newly diagnosed smear-positive (>/=1+ AFB) and whose household contacts are enrolled in the TB-LION study and are receiving nutritional supplementation
* 50 participants will be enrolled and followed for up to 12 months
* Index case and rest of household will receive nutritional supplementation for 6 months
* Stool sample will be collected at the week 1 visit (visit 2)
* Blood samples will be collected at the screening visit, week 1, month 2, and month 6
* Sputum samples will be collected at the screening visit, week 1, week 2, and month 6

LEOPARD Cohort 2-

* Pulmonary TB patients who are newly diagnosed smear-positive (>/=1+ AFB) and whose household contacts are not enrolled in the TB-LION study
* 300 participants will be enrolled and followed for up to 6 months
* Stool sample will be collected at the week 1 visit (visit 2)
* Blood samples will be collected at the screening visit and week 1
* Sputum samples will be collected at the screening visit, week 1, and week 2

ELIGIBILITY:
Inclusion Criteria:

* Sputum Ziehl-Neelsen stain positive for AFB (≥1+)
* Culture or Xpert positive for Mtb; those who are smear+ but ultimately Xpert or culture negative, will be included until their culture results return at which time they will retrospectively be removed from the study.
* No history of TB treatment (i.e., no history of partial or complete treatment for a previous TB episode)
* Has at least 1 household contact with whom they have shared a house with during the previous one month
* Agrees to have household contact notified about study

Exclusion Criteria:

* Household contact ineligible for TB LION study
* Pregnant at enrollment
* Previously diagnosed with diabetes or hemoglobin A1c>6.5% on testing
* No Xpert or culture confirmation and unable to provide sputum sample
* Known multidrug-resistant tuberculosis (MDR) or extensively drug resistant (XDR) TB case at recruitment or found at time of enrollment
* BMI <14 kg/m2
* Lower extremity edema/kwashiorkor
* Reported neuropathy in lower extremities (may result from thiamine deficiency)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is newly diagnosed smear-positive (>/=1+ AFB) pulmonary TB patients living in Puducherry and Tamil Nadu.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2022-04-09 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2025-07-21 (Actual)

PRIMARY OUTCOMES:
Percent of participants who successfully complete TB treatment | 6 months
  The number of participants that successfully completed treatment without bacteriological evidence of failure for two continuous weeks will be divided by the number of participants who started TB treatment.
Body Mass Index (BMI) at the end of treatment | 6 months
  BMI will be calculated as weight/height in kg/m2. The height of participants will be measured by study team members at a home visit . Height will be measured to the nearest 0.5 cm with a stadiometer (or knee height, ulnar length or arm span [demispan] for those persons unable to stand fully erect). Body weight will be measured to the nearest 0.1 kg. Low BMIs <18.5 are associated with malnutrition.
Detection of parasites in stool specimen | 1 week
  Stool specimens collected at the first visit will be tested for intestinal parasites using polymerase chain reaction (PCR).

CONTACTS AND LOCATIONS:
Overall Officials: Pranay Sinha, MD, Principal Investigator — Boston Medical Center; Pakrash Babu Narasimhan, PhD, Principal Investigator — Jawaharlal Institute of Postgraduate Medical Education and Research (JIPMER)
Locations (2):
- Boston Medical Center, Boston, Massachusetts, United States
- Jawaharlal Institute of Postgraduate Medical Education and Research, Puducherry, India

IPD SHARING:
Plan to Share IPD: Undecided